CLINICAL TRIAL: NCT03564314
Title: Strategy for Uptake of Processes for Recognizing and Responding to Acute Kidney Injury
Acronym: SUPPORT AKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other); University of Alberta (Other); Covenant Health, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: REB14-1531
Record Dates: First submitted 2018-05-25; First posted 2018-06-20 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2022-06

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Major surgery; Clinical decision support
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SUPPORT AKI Clinical Decision Support (Experimental): Multidimensional clinical decision support intervention consisting of education and tools to support early recognition and management of AKI, including guidance on fluid therapies, medication management, investigation, and consultation with specialists.
  Interventions: Other: SUPPORT AKI Clinical Decision Support
- Control (No Intervention): Usual care provided to patients with AKI on surgical units.

INTERVENTIONS:
Other: SUPPORT AKI Clinical Decision Support — Surgical units will receive a multidimensional clinical decision support intervention consisting of: (1) electronic and non-computerized tools to alert for early recognition of AKI, (2) educational program for physicians and nursing staff, (3) decision support tools with guidance on fluid therapies, medication management, investigations for AKI, and consultation with specialists.
  Arms: SUPPORT AKI Clinical Decision Support

SUMMARY:
Acute kidney injury (AKI) is common and costly complication of major surgery. AKI can lead to prolonged hospitalization and a higher likelihood of dialysis, chronic kidney disease and death. However, AKI can be reversed when recognized early, by ensuring that patients receive adequate fluids and medications that worsen kidney function or cause toxicity are avoided or appropriately prescribed. Past research suggests that AKI in surgical settings can be missed early in its onset, leading to delayed intervention and progression to more severe stages. The purpose of this project is to implement clinical decision support for early recognition and management of AKI on surgical units in Alberta hospitals, and to determine whether the initiative leads to improvements in the quality of care for AKI, length of hospital stay for patients, and costs to the healthcare system.

DETAILED DESCRIPTION:
Overview: Cluster-randomized stepped-wedge trial to evaluate the impact of implementing a clinical decision support initiative for early recognition and management of hospital-acquired AKI.

Study Population: Adult patients hospitalized on surgical units in Alberta who develop acute kidney injury will be eligible if not already receiving dialysis.

Intervention: The multidimensional clinical decision support intervention consists of: (1) electronic and non-computerized tools for early recognition of AKI, (2) educational program for clinical staff, (3) decision support resources and guidance for the management of AKI and consultation with specialists.

Study Design: Using a stepped-wedge design, eight general and vascular surgery unit clusters in Calgary (Foothills Medical Centre, Peter Lougheed Centre) and Edmonton (University of Alberta Hospital, Grey Nuns Community Hospital), Alberta will be randomly ordered to be sequentially introduced to the clinical decision support intervention. The pre-implementation period will include all patients admitted to the participating hospital units in the year before the random timing of introduction of the initiative on each participating unit. The post-implementation study cohort will include patients admitted in the year after the random timing of introduction of the initiative on each unit. Analysis of processes of care and outcomes will focus on patients on these units who develop AKI during the pre- and post-implementation time periods (i.e. are eligible to receive care under the AKI decision support initiative). Additionally, health care providers (e.g. physicians, nursing staff, pharmacists) who have direct experience with the clinical decision support tools and processes will be invited to participate in the surveys and interviews pre- and post-implementation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age and older) who develop hospital-acquired acute kidney injury on identified general and vascular surgery units in Alberta

Exclusion Criteria:

* Hospitalized on non-surgical units
* Receiving dialysis prior to admission on surgery unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2135 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Progression of AKI | From date of AKI onset to discharge from hospital, assessed up to 30 days
  Incidence of progression of AKI to higher AKI stage (including progression to dialysis or death)

SECONDARY OUTCOMES:
Length of AKI hospital stay, days | From date of AKI onset to discharge from hospital, assessed up to 30 days
  Mean length of hospital stay from acute kidney injury to discharge
Resource use for AKI | Duration of index hospital admission, assessed up to 30 days
  Mean total health care costs of hospital care during the index admission
Time to initial response to AKI | From AKI onset up to 48 hours following AKI onset
  Time from AKI onset to clinical response with fluid or medication management intervention
Volume intervention (change in fluid or diuretic order) for AKI | Within 48 hours following AKI onset
  New or modified intravenous fluid or diuretic order
Adverse medication exposure | Within 48 hours following AKI onset
  Dose modification or suspension or a medication that may cause AKI or that is cleared by the kidney
Medical consultation for AKI | Within 7 days of AKI onset
  Consultation with nephrology or general internal medicine
Change in estimated Glomerular Filtration Rate (eGFR) | From most recent baseline eGFR measurement prior to AKI onset to eGFR measurement closest to 3 months after AKI onset
  The difference in eGFR from baseline to 3 months after development of AKI
Mortality | Within 30 days of AKI onset
  All cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T James, MD, PhD, Principal Investigator — Associate Professor
Locations (4):
- Canada (4):
  - Peter Lougheed Centre, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta